CLINICAL TRIAL: NCT05205993
Title: Investigating the Effectiveness of Innovative Intrauterine Antibiotic Therapy for the Treatment of Patients With Chronic Endometritis
Brief Title: Εffectiveness of Intrauterine Antibiotic Administration for Treatment of Chronic Endometritis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Genesis Athens Clinic (Other)
Collaborators: National and Kapodistrian University of Athens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IAI-1
Record Dates: First submitted 2021-12-23; First posted 2022-01-25 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Chronic Endometritis
MeSH Terms: interventions — Administration, Oral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intrauterine infusion of antibiotics (Experimental): Thirty women will receive only intrauterine infusion of antibiotics for 30 days.
  Interventions: Drug: Intrauterine infusion
- Combination of intrauterine infusion and oral administration of antibiotics (Experimental): Thirty women will receive a combination of intrauterine infusion and oral administration of antibiotics for 30 days.
  Interventions: Drug: Intrauterine infusion; Drug: Oral administration
- Oral administration of antibiotics (Active Comparator): Thirty women will receive only oral administration of antibiotics for 30 days.
  Interventions: Drug: Oral administration

INTERVENTIONS:
Drug: Intrauterine infusion — A total of 10 intrauterine infusions of 3ml of ciprofloxacin at a concentration of 200 mg/100 ml
  Arms: Combination of intrauterine infusion and oral administration of antibiotics; Intrauterine infusion of antibiotics
Drug: Oral administration — per os antibiotic administration as the standard line of strategy for treating CE of doxycycline at a dosage of 100mg twice a day and metronidazole of 500mg twice a day for a total of 30 days
  Arms: Combination of intrauterine infusion and oral administration of antibiotics; Oral administration of antibiotics

SUMMARY:
Chronic Endometritis (CE) is related to infertility and entails a challenging management. This study investigates the treatment of off-label intrauterine antibiotic infusion either separately or combined with oral antibiotic administration, and it assesses respective performance against the gold standard treatment of oral antibiotic adminstration. Data sourced herein reports on treatment efficiency, defined as a negative diagnosis for chronic endometritis.

DETAILED DESCRIPTION:
An infectious endometrial environment caused by certain pathologies could compromise establishment of the initial interaction between the embryo and the endometrium. Chronic endometritis (CE) is a case of a persistent endometrial inflammation caused by infectious agents namely Escherichia Coli, Enterococcus faecalis, Streptococcus agalactiae, Mycoplasma, Ureaplasma, and Chlamydia. The perplexity of managing CE is attributed to its asymptomatic nature rendering a definitive diagnosis rather challenging. The list of potential symptoms is limited and vague while manifestation of the disease may be mild and may not correspond to severity. Symptoms include pain in the pelvic cavity, dispareunia, uterine bleeding, vaginal infections and cystitis, and mild gastro-intestinal discomfort. CE is described as a chronic disorder due to its long duration and persistent nature, with potentially slow progression and complex causality, severely compromising reproductive potential of patients.

The antibiotic treatments are primarily administered orally and endometrial re-examination is performed following treatment. It should be emphasized that apart from the differences in the types of antibiotics included, there are also significant discrepancies regarding the dosage of each antibiotic and the different schemes suggested by each practice. Following the antibiotic regime, endometrial receptivity is anticipated to improve. However, a significant correlation between the antibiotic therapeutic approach and a positive results in IVF has failed to be established in literature, indicating that oral antibiotic administration is unseccessful in improving IVF outcome.

A pilot study published by the investigators indicated that combination of intrauterine infusion of antibiotics and oral administration can be more effective in treating CE than solely oral administration. However, it has not been evaluated if sole intrauterine infusion of antibiotics can be of similar effectiveness when compared to the combined regime including intrauterine infusion and oral andministration, or when compared to the gold standard treatment including only oral administration of antibiotics.

ELIGIBILITY:
Inclusion Criteria:

* Positive diagnosis of CE following hysteroscopy and endometrial biopsy (positive diagnosis is required by both evaluations)
* Signed Informed Consent
* 18.5 < BMI < 30

Exclusion Criteria:

* Diagnosed endometriosis or other related Pelvic Inflammatory Disorder (PID)
* Current or previous cancer diagnosis
* Auto-immune or genetic disorders
* Menstrual cycle disorders

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-01-19 (Actual); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Negative diagnosis of CE following hysteroscopy and endometrial biopsy | Negative diagnosis of CE will be assessed in one month -immidiately after treatment completion-.
  All participants will be subjected to hysteroscopy and endometrial biopsy following completion of treatment. Regarding hysteroscopy the presence of endometritis will be evaluated according to the published unified diagnostic criteria for CE. The endometrial biopsy will be performed employing a pipelle. To minimize contamination risk, following the placement of a vaginal speculum and cleaning external uterine ostium with an iodine solution, the pipelle will be inserted under visual control into the uterine cavity ensuring avoidance of any contact with vaginal walls. Endometrial samples will be diluted into 2 ml of saline for histological analysis. For histological analysis the endometrium samples will be fixated employing neutral formalin and paraffin. To stain the microsections, hematoxyline and eosin will be engaged. CD138 staining will be performed and positivity will indicate a CE diagnosis (>1 plasma cell per 10HPFs). A negative CE diagnosis should be confirmed by both assessments

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v6.0 | Side-effects will be monitored for one month from treatment initiation which is until completion of treatment
  Number of reports of side-effects according to CTCAE v6.0 per treated patients

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Sfakianoudis, MD, Principal Investigator — Genesis Athens Clinic
Locations (1):
- Genesis AC, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pantos K, Simopoulou M, Maziotis E, Rapani A, Grigoriadis S, Tsioulou P, Giannelou P, Nitsos N, Tzonis P, Koutsilieris M, Sfakianoudis K. Introducing intrauterine antibiotic infusion as a novel approach in effectively treating chronic endometritis and restoring reproductive dynamics: a randomized pilot study. Sci Rep. 2021 Aug 2;11(1):15581. doi: 10.1038/s41598-021-95072-w. PMID 34341409